CLINICAL TRIAL: NCT07275112
Title: Cross-cultural Adaptation of the TENDINopathy Severity Assessment-Achilles (TENDINS-A) for the Spanish Population and Evaluation of Its Reliability and Validity in Accordance With COSMIN Recommendations
Brief Title: Cross-cultural an Reliability and Validity Evaluation of TENDINS-A in Spain
Status: Completed | Type: Observational
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, SERGIO MONTERO NAVARRO, Principal Investigator, Cardenal Herrera University
Other Study IDs: CEEI 24/558
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Achilles Tendinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cross-cultural adaptation — Cultural and linguistic adaptation process including forward/back translation, expert review, and cognitive debriefing and forward translation, back-translation, expert panel evaluation, cognitive interviews.
Other: Evaluation of reliability and validity — Administration of adapted instrument for reliability and validity assessment and psychometric testing of the adapted questionnaire to evaluate reliability and validity.

SUMMARY:
Volunteers who want to participate in the study will read the general information of the study and sign the informed consent to participate in the study.

Once the informed consent has been read and delivered, the evaluator will check that they meet the inclusion criteria. After the data collection, a randomization (Epidat V4.0) of the selected subjects will be carried out to assign them to one of the intervention groups.

Patients must present Achilles pathology and will be recruited through a network of physiotherapy clinics distributed across Spain.

The physiotherapist responsible for their treatment will invite them to participate in the study by providing a QR code granting access to all relevant study documentation. This documentation will include a checkbox in which the patient must indicate that, after reading all the pertinent information, they consent to participate. Without this explicit consent, marked via the checkbox, participation will not be possible.

Once consent is provided, the patient will gain access to three questionnaires to be completed at the same time: VISA-A, FAOS, and TENDINS-A. After 48 hours, they will receive a link to complete the TENDINS-A retest.

When the participant has completed all four questionnaires (VISA-A, FAOS, TENDINS-A, and the TENDINS-A retest), their participation in the study will be considered complete.

The sample size will be calculated following COSMIN recommendations, aiming for a minimum of more than 100 participants to ensure excellent reliability.

ELIGIBILITY:
Inclusion Criteria:

* Present Achilles tendinopathy
* Accept participation in the study (acceptance of informed consent)
* Being a native Spanish speaker
* Be in an age range between 18 and 55 years.
* Do not present any exclusion criteria.

Exclusion Criteria:

* Complete or partial tendon rupture
* Other recent injuries in the affected limb
* Previous surgery in the limb
* Haglund syndrome
* Inflammatory diseases
* Autoimmune diseases

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with Achilles tendinopathy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2025-12-05 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-19 (Actual)

PRIMARY OUTCOMES:
Test-retest reliability (Intraclass Correlation Coefficient (ICC 2,1)). | Baseline and 2-3 days after the first administration.
  Degree of stability of the adapted questionnaire scores when administered twice to the same participants under similar conditions. ICC values with 95% confidence intervals.
Internal consistency (Cronbach's alpha coefficient; ranges from 0 to 1.). | At baseline.
  Internal homogeneity of the items of the adapted questionnaire. Calculation of Cronbach's alpha for total score and subscales (if applicable). 0.90 or higher: Excellent reliability.
  0.80 to 0.89: Good internal consistency. 0.70 to 0.79: Acceptable reliability (the minimum standard in research). Less than 0.50: Unacceptable consistency.
Construct validity | At baseline.
  Degree to which the adapted instrument reflects the theoretical construct it is intended to measure. Exploratory Factor Analysis (EFA) and/or Confirmatory Factor Analysis (CFA), depending on design.

SECONDARY OUTCOMES:
Age (years) | At baseline.
Sex (Male and female) | At baseline.
Weight (kg) | At baseline.
BMI (body max index kg/cm2) | At baseline.
Height (cm) | At baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad CEU Cardenal Herrera, Elche, Alicante, Spain

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-11-28): https://cdn.clinicaltrials.gov/large-docs/12/NCT07275112/Prot_SAP_ICF_000.pdf